CLINICAL TRIAL: NCT03830814
Title: What Are the Effects of Sacubitril/Valsartan on the Heart Functions? Can It Increase the Ejection Fraction?
Brief Title: The Effects of Sacubitril/Valsartan on the Heart Functions
Status: Completed | Type: Observational
Sponsor: The Young Investigator Group of Cardiovascular Research (Network)
Responsible Party: Sponsor
Other Study IDs: YIG01201901
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Drug Effect
Keywords: Sacubitril/Valsartan; Heart Failure; Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cases: Patients with heart failure with reduced ejection fraction (HRrEF) who have indications for the use of sacubitril/valsartan as recommended by recent guidelines
  Interventions: Procedure: Echocardiography

INTERVENTIONS:
Procedure: Echocardiography — Basal two dimensional and three dimensional echocardiographic parameters were compared to those obtained 3 months after starting the sacubitril/valsartan treatment

SUMMARY:
Background:

Sacubitril/valsartan, has been found to be more beneficial than enalapril for reducing the incidences of sudden cardiac death, death from worsening heart failure (HF), and hospitalization. However, there is no prospective echocardiographic data describing the effects of sacubitril/valsartan on the heart functions and left ventricular (LV) reverse remodeling. Therefore, the aim of our study was to evaluate the effects of sacubitril/valsartan on the LV functions using two dimensional (2D), three dimensional (3D) echocardiography and the 3D strain parameters.

Methods:

In 100 patients with HF with reduced ejection fraction (HRrEF) who have indications for the use of sacubitril/valsartan as recommended by recent guidelines were prospectively enrolled. The basal 2D and 3D echocardiographic parameters were compared to those obtained 3 months after starting the sacubitril/valsartan treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age is more than or equal 18 years old
* Able to provide written informed consent
* Indicated for the use of sacubitril/valsartan as recommended by the European Society of Cardiology (ESC) heart failure guidelines 2016
* Left ventricular ejection fraction of 40% or less

Exclusion Criteria:

* Cardiac resynchronization therapy (CRT) device implantation less than 3 months prior to the start of this study or CRT implantation intentions
* Atrial fibrillation
* Poor echocardiographic images
* Sacubitril/valsartan treatment intolerance during the follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred patients with heart failure with reduced ejection fraction (HRrEF) who have indications for the use of sacubitril/valsartan as recommended by recent guidelines were prospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Two dimensional left ventricular ejection fraction | 3 months
  Two dimensional ejection fraction is measured as baseline and after 3 months follow-up
Three dimensional left ventricular ejection fraction | 3 months
  Three dimensional ejection fraction is measured as baseline and after 3 months follow-up

SECONDARY OUTCOMES:
Two dimensional left ventricular volumes | 3 months
  Two dimensional left ventricular volumes are measured as baseline and after 3 months follow-up
Three dimensional left ventricular volumes | 3 months
  Three dimensional left ventricular volumes are measured as baseline and after 3 months follow-up